CLINICAL TRIAL: NCT02011659
Title: A Randomized Prospective Study of Scheduled Intravenous Ramosetron for the Prevention of Nausea and Vomiting in Hospitalized Patients After Gynecologic Laparoscopy
Brief Title: Long Term Prevention of Nausea and Vomiting in Gynecologic Laparoscopy
Acronym: PONV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Insurance Service Ilsan Hospital (Other)
Responsible Party: Principal Investigator, San-Hui Lee, Clinical assistant professor, National Health Insurance Service Ilsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PONV-NHIS-GYN-001
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Uterine Myoma, Ovary Neoplasm, Adenomyosis
Keywords: Ramosetron, postoperative nausea and vomiting, laparoscopy
MeSH Terms: conditions — Myofibroma; Ovarian Neoplasms; Adenomyosis; Postoperative Nausea and Vomiting; Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ramosetron (Active Comparator)
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron

SUMMARY:
To compare postoperative nausea and vomiting (PONV) and perioperative outcomes of gynecologic patients undergoing laparoscopic surgery after scheduled administration of intravenous Ramosetron during hospital stays.

* Randomized controlled arm : Placebo versus Ramosetron injection
* Administration schedule : immediate postoperative status, 12 hrs after surgery, 36hrs after surgery

DETAILED DESCRIPTION:
Surgical outcomes including operative time, blood loss, Hb change, postoperative pain, nausea/vomiting scale, times of rescue therapy, and complications

ELIGIBILITY:
Inclusion Criteria:

* Age: 18< or =, = or <70 with benign gynecologic disease
* ASA-Class I-II
* No-definite malignancy by US, CT/MRI, CA 125 < 500IU/ml
* Non-smoker

Exclusion Criteria:

* Conversion to laparotomy
* Hx of malignancy
* Smoker
* Suspicious malignancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Incidence or intensity of PONV | during postoperative hospital stays (2 days)

SECONDARY OUTCOMES:
Adverse reaction associated with Ramosetron injection | Postoperatvie 7 days (at OPD based)

CONTACTS AND LOCATIONS:
Locations (1):
- National Health Insurance Service Ilsan Hospital, Goyang-si, South Korea

REFERENCES:
- [Derived] Li SC, Wang Y, Choi SJ, Jung YS, Han KH, Chung IB, Lee SH. Scheduled injection of ramosetron for prevention of nausea and vomiting following single-port access total laparoscopic hysterectomy: a prospective randomized study. Obstet Gynecol Sci. 2019 Sep;62(5):344-351. doi: 10.5468/ogs.2019.62.5.344. Epub 2019 Jul 23. PMID 31538078